CLINICAL TRIAL: NCT02821052
Title: Post-marketing Surveillance (Special Use-results Surveillance) on Long-term Use With Ryzodeg®.
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN5401-4152; U1111-1149-9518 (Other: WHO)
Record Dates: First submitted 2016-06-29; First posted 2016-07-01 (Estimated); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — insulin degludec, insulin aspart drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- insulin degludec/insulin aspart
  Interventions: Drug: insulin degludec/insulin aspart

INTERVENTIONS:
Drug: insulin degludec/insulin aspart — Enrolled patients will be treated with Ryzodeg® under routine clinical practice.

SUMMARY:
This trial is conducted in Asia. The aim of this Non-interventional study is to investigate the long-term safety and effectiveness of Ryzodeg® (insulin degludec/insulin aspart) in Japanese patients with diabetes mellitus requiring insulin therapy under normal clinical practice conditions.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol)
* The decision to initiate treatment with commercially available Ryzodeg® has been made by the patient/Legally Acceptable Representative (LAR) and the treating physician before and independently from the decision to include the patient in this study
* Patients with diabetes mellitus requiring insulin therapy for whom the physician has decided to start treatment with Ryzodeg®
* Male or female, no age limitation

Exclusion Criteria:

* Patients who are or have previously been treated with Ryzodeg®
* Previous participation in this study. Participation is defined as having given informed consent in this study
* Patients with a history of hypersensitivity to study product components
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Japanese patients with diabetes mellitus requiring insulin therapy under normal clinical practice conditions.
Sampling Method: Non-Probability Sample
Enrollment: 1355 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2018-11-24 (Actual); Study Completion 2018-11-24 (Actual)

PRIMARY OUTCOMES:
Incidence of AEs (adverse event) | Year 0-1

SECONDARY OUTCOMES:
Incidence of SADRs (Serious Adverse Drug Reactions) | Year 0-1
Severe hypoglycaemic episodes | Year 0-1
Incidence of Serious allergic reactions (systemic or localized, including injection site reactions) | Year 0-1
Change in Glycosylated haemoglobin A1c (HbA1c) | Week 0, week 52

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Tokyo, Japan

REFERENCES:
- [Derived] Katabami T, Eriksen KT, Yamamoto Y, Ishigaki Y. Long-Term Safety and Clinical Outcomes with Insulin Degludec/Insulin Aspart Treatment in Japanese Patients with Diabetes: A Real-World, Prospective, Observational Study. Adv Ther. 2022 Jan;39(1):544-561. doi: 10.1007/s12325-021-01978-2. Epub 2021 Nov 20. PMID 34800283
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com